CLINICAL TRIAL: NCT02868983
Title: Integrating Behavioral Health and Primary Care for Comorbid Behavioral and Medical Problems
Acronym: IBHPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Collaborators: Arizona State University (Other); State University of New York at Buffalo (Other); Case Western Reserve University (Other); DARTNet (Unknown); National Committee for Quality Assurance (Other); University of Massachusetts, Worcester (Other); Patient Centered Outcomes Oriented Research Institute (Unknown)
Responsible Party: Principal Investigator, Benjamin Littenberg, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: WLPS-1409-24372
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Arthritis; Asthma; Chronic Obstructive Lung Disease; Diabetes; Heart Failure; Hypertension; Anxiety; Chronic Pain; Depression; Fibromyalgia; Insomnia; Irritable Bowel Syndrome; Problem Drinking; Substance Use Disorder
MeSH Terms: conditions — Arthritis; Asthma; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Heart Failure; Hypertension; Anxiety Disorders; Chronic Pain; Depression; Fibromyalgia; Sleep Initiation and Maintenance Disorders; Irritable Bowel Syndrome; Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integration (Experimental): The intervention consists of training for practice leaders, BHCs, PCPs, and office staff, a Protocolized Redesign Process support for practice redesign, and a toolkit of suggested tactics for implementing Tasks A through D:
  A. Identification B. Assessment C. Treatment D. Surveillance
  Interventions: Other: Integration
- Co-Location (No Intervention): A Behavioral Health Clinician (BHC) such as a psychologist or counselor is housed in or near the primary care practice.

INTERVENTIONS:
Other: Integration — The intervention consists of training for practice leaders, BHCs, PCPs, and office staff, a Protocolized Redesign Process support for practice redesign, and a toolkit of suggested tactics for implementing Tasks A through D:
  A. Identification B. Assessment C. Treatment D. Surveillance
  Arms: Integration

SUMMARY:
Behavioral problems are part of many of the chronic diseases that cause the majority of illness, disability and death. Tobacco, diet, physical inactivity, alcohol, drug abuse, failure to take treatment, sleep problems, anxiety, depression, and stress are major issues, especially when chronic medical problems such as heart disease, lung disease, diabetes, or kidney disease are also present. These behavioral problems can often be helped, but the current health care system doesn't do a good job of getting the right care to these patients.

Behavioral health includes mental health care, substance abuse care, health behavior change, and attention to family and other psychological and social factors. Many people with behavioral health needs present to primary care and may be referred to mental health or substance abuse specialists, but this method is often unacceptable to patients. Two newer ways have been proposed for helping these patients. In co-location, a behavioral health clinician (such as a Psychologist or Social Worker) is located in or near the primary practice to increase the chance that the patient will make it to treatment. In Integrated Behavioral Health (IBH), a Behavioral Health Clinician is specially trained to work closely with the medical provider as a full member of the primary treatment team.

The research question is: Does increased integration of evidence-supported behavioral health and primary care services, compared to simple co-location of providers, improve outcomes? The key decision affected by the research is at the practice level: whether and how to use behavioral health services.

The investigators plan to do a randomized, parallel group clustered study of 3,000 subjects in 40 practices with co-located behavioral health services. Practices randomized to the active intervention will convert to IBH using a practice improvement method that has helped in other settings. The investigators will measure the health status of patients in each practice before and after they start using IBH. The investigators will compare the change in those outcomes to health status changes of patients in practices who have not yet started using IBH.

The investigators plan to study adults who have both medical and behavioral problems, and get their care in Family Medicine clinics, General Internal Medicine practices, and Community Health Centers.

DETAILED DESCRIPTION:
The chronic diseases that drive the majority of mortality, morbidity and cost in America and around the globe are largely behavioral in origin or management. Tobacco, diet, physical inactivity, alcohol, substance abuse, non-adherence to treatment, insomnia, anxiety, depression, and stress are major causes of morbidity, mortality and expense, especially when chronic medical problems such as heart disease, lung disease, diabetes, or arthritis are also present. Behavioral problems can often be effectively managed with improved outcomes for patients, their families and the health care system, but the current health care system is often unable to provide such care.

Behavioral Health includes mental health care, substance abuse care, health behavior change, and attention to family and other psychosocial factors. Many people with behavioral health needs present to primary care and may be referred to mental health or substance abuse specialists, but this method is often unacceptable to patients. Two newer models have been proposed for helping these patients. In co-location, a behavioral health provider is located in or near the primary practice to increase the likelihood of successful referral and treatment initiation. An alternative is Integrated Behavioral Health (IBH) in which a Behavioral Health Clinician is specially trained to work closely with the medical provider as a full member of the primary treatment team. Although it is clear that the status quo of under-diagnosis or inadequate referral and treatment is not acceptable, it is not known which of the alternative models is best.

The research question is: Does increased integration of evidence-supported behavioral health and primary care services, compared to simple co-location of providers, improve patient-centered outcomes in patients with multiple morbidities? The key health decisions affected by the research are those made at the practice level: whether and how best to incorporate behavioral health (BH) services. At the patient level, the decision of whether to seek out or accept offered BH services will be influenced by the manner they are made available.

Aim 1: Determine if increased integration of evidence-supported behavioral health and primary care results in better patient-centered outcomes than simple co-location of behavioral providers without systematic integration.

Aim 2: Determine if structured improvement process techniques are effective in increasing BH integration.

Aim 3: Explore how contextual factors affect the implementation and patient centeredness of integrated BH care.

Aim 4: Assess the costs of implementing integration in this setting.

Aim 5: Covid Enhancement: What is the effect of the pandemic upon the effectiveness of IBH?

This is a prospective, cluster-randomized, mixed methods comparison of co-location of BH services vs. IBH in 3,000 subjects in 40 primary care practices around the US.

Usual care (the control comparator) for practices attempting to deliver BH services is co-location of a BH clinician within or adjacent to the primary care facility, without increased integration. The active comparator (the intervention) is Integrated Behavioral Health to support the delivery of protocol supported, stepped, data-driven, evidence-supported, BH care. In both cases, the expenses (such as salaries for the Behavioral Health Clinicians) will be paid by the practices. The intervention consists of training for practice leaders, Behavioral Health Clinicians, primary care providers, and office staff, a Structured Improvement Process support for practice redesign, and a toolkit of suggested tactics for implementing BH.

The target patient population is adults with multiple comorbid medical and behavioral problems receiving services in the target practice settings: Family Medicine clinics, General Internal Medicine practices, and Community Health Centers. The investigators will enroll 40 practices from around the country to represent a broad spectrum of US primary care sites including those serving racial and ethnic minority groups, low-income groups, women, seniors, residents of rural areas, and patients with special health needs, disabilities, multiple chronic diseases, low health literacy or numeracy and/or limited English proficiency. The intervention will be directed at the practices and its impact measured in a randomly selected sample of 75 patients with behavioral health needs from each practice for a total of 3000 patients followed for 2 years.

The primary outcome is the PROMIS-29, a patient-centered measure of global health and functioning. Secondary analyses will assess other outcomes important to patients as well subgroup analyses to allow exploration of what types of patients and practices benefit most from Integrated Behavioral Health. Aim 2 will study the effect of the intervention on practice structure and processes. Aim 3 will identify barriers and supports for successful integration. Aim 4 will assess costs of implementation.

The analyses for Aims 1 and 2 will use generalized linear mixed models of patient health status to perform intention-to-treat analyses as a function of experimental condition (co-location vs. integration), patient characteristics, and time of measurement, with multiple measures clustered within patients and patients clustered within practices. The parameters of interest are the central tendency (mean), statistical significance (P values) and 95% confidence intervals (CI) of the adjusted change in PROMIS-29 domain score since before the intervention. Each of the 8 outcome domains in the PROMIS-29 will be modeled individually as 8 separate hypotheses with adjustment for multiple comparisons. Secondary outcomes (Communication, Empathy, Adherence, etc.) will use similar models. Aim 3 will use mixed methods analysis of surveys, focus groups, key informant interviews and other data sources to explore the relationship between the context of the intervention and the patient-centeredness of the resultant care. Aim 4 will use a survey of practice managers in a subset of practices to collect information on staffing changes,staff time, supplies and capital expenses incurred as part of implementation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* At least one target chronic medical condition:
* arthritis
* asthma
* chronic obstructive lung disease
* diabetes
* heart failure
* or hypertension.
* Evidence of a behavioral problem or need:
* Diagnosis of:
* anxiety
* chronic pain including headache
* depression
* fibromyalgia
* insomnia
* irritable bowel syndrome
* problem drinking
* substance use disorder
* OR persistent use of certain medications used for behavioral concerns:
* antidepressants
* anxiolytics
* opioids
* antineuropathy agents
* OR persistent failure to attain physiologic control of a medical problem:
* blood pressure>165 while on 3 or more medications
* A1C > 9% for 6 months)
* OR the presence of three or more of the target chronic medical conditions.

Exclusion Criteria:

* Not seeking care at a participating practice
* Inability to consent due to cognitive and/or developmental impairment/delays
* Living in the same household as a previously enrolled study participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4025 (Actual)
Dates: Start 2016-04; Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
PROMIS-29 v2 | 24 months
  Change in general health

SECONDARY OUTCOMES:
CAHPS 12-Month PCMH Adult Questionnaire 2.0 | 24 months
  Quality of provider communication
Consultation and Relational Empathy measure | 24 months
  Quality of provider empathy
Patient Activation Measure-13 | 24 months
  Self-management
Modified Self-reported Medication-taking Scale | 24 months
  Medication adherence
Patient Report of Utilization | 24 months
  Health care utilization
Restricted Activity Days | 24 months
  Time lost due to disability
Duke Activity Status Index | 24 months
  Physical Function
Hgb A1C | 24 months
  Glycemic control
30-day use | 24 months
  Substance Use disorder & Problem Drinking
Global Appraisal of Individual Needs - Short Screener | 24 months
  Substance Use disorder & Problem Drinking
Systolic blood pressure | 24 months
  Hypertension
Asthma Symptom Utility Index | 24 months
  Asthma symptoms

OTHER OUTCOMES:
Staff Burnout | 24 months
  Ancillary study: What is the effect of the IBH-PC intervention on staff burnout?
Practice Integration Profile | 24 months
  Aim 2: Self-report by practice staff on degree of integration of behavioral and medical services
Costs of Implementation | 24 months
  Aim 4: Staff time, supplies, capital and other expenses
Patient Centeredness Index | 24 months
  Patient-report of patient-centeredness of their Primary Care practice
Covid-19 practice measures | 24-32 months
  Impact of Covid-19 at the practice level
Covid-19 patient measures | 24-32 months
  Impact of Covid-19 at the patient level

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Littenberg, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete, cleaned, de-identified copy of the final dataset used in conducting the final analyses will be made available within one year after the completion of the study. It will include a data dictionary with response and missing values defined as well as a complete set of survey instruments (excluding copyright protected material not licensed for transfer). The data will be available as an encrypted Stata data set or comma-separated file. The investigators will not make data from qualitative results available because of the potential for identifying individuals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after study completion for at least one year.
Access Criteria: All requests will be reviewed by the project's Ancillary Studies committee to ensure scientific validity and lack of overlap with ongoing analyses.

REFERENCES:
- [Derived] van Eeghen C, Soucie J, Clifton J, Hitt J, Mollis B, Rose GL, Scholle SH, Stephens KA, Zhou X, Baldwin LM. Implementation outcomes from a randomized, controlled trial of a strategy to improve integration of behavioral health and primary care services. BMC Health Serv Res. 2024 Nov 8;24(1):1361. doi: 10.1186/s12913-024-11801-7. PMID 39511571
- [Derived] Nagykaldi Z, Littenberg B, Bonnell L, Breshears R, Clifton J, Crocker A, Hitt J, Kessler R, Mollis B, Miyamoto RES, van Eeghen C. Econometric evaluation of implementing a behavioral health integration intervention in primary care settings. Transl Behav Med. 2023 Aug 11;13(8):571-580. doi: 10.1093/tbm/ibad013. PMID 37000706
- [Derived] Rose GL, Bonnell LN, Clifton J, Natkin LW, Hitt JR, O'Rourke-Lavoie J. Outcomes of Delay of Care After the Onset of COVID-19 for Patients Managing Multiple Chronic Conditions. J Am Board Fam Med. 2022 Dec 23;35(6):1081-1091. doi: 10.3122/jabfm.2022.220112R1. Epub 2022 Nov 17. PMID 36396416
- [Derived] Bonnell LN, Troy AR, Littenberg B. Exploring non-linear relationships between neighbourhood walkability and health: a cross-sectional study among US primary care patients with chronic conditions. BMJ Open. 2022 Aug 19;12(8):e061086. doi: 10.1136/bmjopen-2022-061086. PMID 35985786
- [Derived] Ma KPK, Mollis BL, Rolfes J, Au M, Crocker A, Scholle SH, Kessler R, Baldwin LM, Stephens KA. Payment strategies for behavioral health integration in hospital-affiliated and non-hospital-affiliated primary care practices. Transl Behav Med. 2022 Aug 17;12(8):878-883. doi: 10.1093/tbm/ibac053. PMID 35880768
- [Derived] Cross AJ, Thomas D, Liang J, Abramson MJ, George J, Zairina E. Educational interventions for health professionals managing chronic obstructive pulmonary disease in primary care. Cochrane Database Syst Rev. 2022 May 6;5(5):CD012652. doi: 10.1002/14651858.CD012652.pub2. PMID 35514131
- [Derived] van Eeghen C, Hitt JR, Pomeroy DJ, Reynolds P, Rose GL, O'Rourke Lavoie J. Co-creating the Patient Partner Guide by a Multiple Chronic Conditions Team of Patients, Clinicians, and Researchers: Observational Report. J Gen Intern Med. 2022 Apr;37(Suppl 1):73-79. doi: 10.1007/s11606-021-07308-0. Epub 2022 Mar 29. PMID 35349025
- [Derived] Crocker AM, Kessler R, van Eeghen C, Bonnell LN, Breshears RE, Callas P, Clifton J, Elder W, Fox C, Frisbie S, Hitt J, Jewiss J, Kathol R, Clark/Keefe K, O'Rourke-Lavoie J, Leibowitz GS, Macchi CR, McGovern M, Mollis B, Mullin DJ, Nagykaldi Z, Natkin LW, Pace W, Pinckney RG, Pomeroy D, Pond A, Postupack R, Reynolds P, Rose GL, Scholle SH, Sieber WJ, Stancin T, Stange KC, Stephens KA, Teng K, Waddell EN, Littenberg B. Integrating Behavioral Health and Primary Care (IBH-PC) to improve patient-centered outcomes in adults with multiple chronic medical and behavioral health conditions: study protocol for a pragmatic cluster-randomized control trial. Trials. 2021 Mar 10;22(1):200. doi: 10.1186/s13063-021-05133-8. PMID 33691772